CLINICAL TRIAL: NCT05474066
Title: Pilot Trial Examining the Impact of Training Related Sub-Concussive Forces On Cognition and Selected Electroencephalogram Measures In Canadian Special Forces Members
Brief Title: ERP Changes Pre and Post Military Changes
Status: Recruiting | Type: Observational
Sponsor: Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Principal Investigator, Gaurav Gupta, Co Investigator, Canadian Forces Health Services Centre Ottawa
Other Study IDs: 2022-016
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Brain Concussion
Keywords: erp; eeg; military
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pre and Post Training: A sample will be recruited from a group of 20 CAF SOF personnel ages 18-65 will be assessed twice: pre and post-special forces military training. All members enrolled in this training will be invited to participate in the study. Testing periods will be about 4 weeks apart, with post training testing within 1 week of conclusion of the exercise. Patients will be recruited from within the Canadian Special Operation Forces community. Recruitment and study will take place starting in September 2022 and continue until complete which is estimated to be approximately 12 months. Participants will be made aware of the study through recruitment letter sent as part of their training package (Appendix A). They will be allowed questions prior to enrollment or at any point during participation.
  Interventions: Device: ERP Testing

INTERVENTIONS:
Device: ERP Testing — * Attention & Concentration:
  * Continuous Visual Memory Test (CVMT):
  * Flanker Task:
  * Hayling Test:

SUMMARY:
This study looks to investigate the cognitive effects associated with intense, military combat training regimens or so-called repetitive sub-concussive forces. Specifically, study participants will undergo cognitive testing in tandem with EEG recordings pre- and post-military training to assess cognition.

DETAILED DESCRIPTION:
Background Despite the high prevalence of cognitive issues in Veterans and active military personnel, there is relatively little understanding regarding the cognitive effects following intense, military training regimens designed to reflect a combat environment and blast exposure. Anecdotal evidence has shown that soldiers complain of cognitive issues post-training similar to those who have sustained brain trauma. Accordingly, this study looks to investigate the cognitive effects associated with intense, military combat training regimens or so-called repetitive sub-concussive forces. Specifically, study participants will undergo cognitive testing in tandem with EEG recordings pre- and post-military training to assess cognition.

Research Objective To assess the effects of repetitive, sub-concussive exposure (RSCE) on cognitive functioning and brain electrophysiology in Special Operation Forces (SOF) personnel. Furthermore, the relation between repetitive sub-concussive exposure and symptoms will be clarified.

Participants and Procedure 20 SOF members will complete a symptom profile, a vestibular ocular motor screening (VOMS), ImPACTTM Cognitive Testing and VoxNeuroTM Electroencephalogram (EEG) assessment pre-and post-training to assess cognitive functioning in the following domains: attention and concentration, working memory, and information processing. Investigators will look for correlations pre and post training

The cognitive assessment(s) to be taken are:

1. ImPact Cognitive Testing
2. VoxNeuro Assessment (EEG)

   1. Attention & Concentration Test - 10min
   2. Continuous Visual Memory Test - 5min
   3. Flanker Test (Optional) - 10min
   4. Hayling Test (TBD - Currently only an English version available) - 10min

      Test Descriptions
      * Participants will keep logbooks looking at trauma exposure to help identify occupational vs non occupational causes, however given the intensity and length of the course significant non Paroccupational exposure is unlikely.
      * Blast Measurement will be monitored using a validated system of three worn blast gauges (Black-box Biometrics Inc.). These gauges - placed on the back of the helmet, non-firing shoulder, and chest - will be used to collect blast overpressure exposure levels above 0.5 psi at the location of the participant during the breaching events. Blast gauges will be issued to all participants prior to blast overpressure exposure and monitored throughout the duration of the study.
      * Vestibular Ocular Motor Screening (VOMS) consists of symptom reporting (eg headache, dizziness, nausea, and fogginess) ranging from 0 (none) to 10 (severe) after testing smooth pursuits, saccades (horizontal and vertical), convergence, Neer Point of Convergence (NPC) distance, horizontal VOR, vertical VOR, and visual motor sensitivity (VMS). For the purpose of this study, we will use the VOMS cutoff scores of ≥2 total symptom score on any VOMS subscale and/or ≥5 cm on NPC average distance
      * ImPACT is an FDA cleared online tool for baseline and post-injury testing. It measures patient reported symptoms, visual and verbal memory, reaction time, and processing speed to help determine if a patient can safely return to activity.
      * VoxNeuro Assessment:

        * Attention & Concentration: An auditory oddball task where the participant is asked to identify the difference between one (1) or more auditory stimuli while EEG is recorded simultaneously to assess Attention and Concentration function at the neurophysiological level.
        * Continuous Visual Memory Test (CVMT): A visual task whereby participants are asked to differentiate between visual stimuli that have been previously presented to them and newly presented visual stimuli while EEG is recorded simultaneously to assess Memory function at the neurophysiological level.
        * Flanker Task: This test consists of participants identifying target stimulus while a target is flanked by non-target stimuli which correspond either to the same directional response as the target (congruent flankers), to the opposite response (incongruent flankers), or to neither (neutral flankers). The test is administered while EEG is recorded simultaneously to assess Executive Function and Response Inhibition at the neurophysiological level.
        * Hayling Test: This test consists of participants being aurally presented congruent and incongruent sentences; whereby, the congruent sentences are "normal" sentences with the final word being correct (e.g., "The pizza was too hot to eat"). In contrast, the incongruent sentences have the final word of a sentence being incorrect (e.g., The pizza was too hot to sing"). The test is administered while EEG is recorded simultaneously to assess Language Comprehension at the neurophysiological level.

      Biological Markers Measured (up to 7) ● N100/P200 - Auditory and Visual Processing
      * N100 ERP is a temporal and frontal component elicited by auditory stimuli. The response is associated with perception.
      * P200 ERP is mainly exhibited at the frontal and occipital lobes and represents higher order perceptual processes such as visual search, language, context information, memory and repetition effects. I.e. all processes modulated by attention.

        * N200 - Information Processing and Executive Function
      * N200 is a centro-cortical component associated with conscious stimuli detection (i.e. information processing and response inhibition) ● P300 - Attention and Memory
      * The P3a is a fronto-central component associated with attention orienting and is followed by the P3b, a centro-parietal component often linked to processes related to memory and attention allocation

        ● N400 - Language Comprehension (TBD)
      * N400 is a central component and acts as the normal brain response to semantic stimuli. For example, words, sign language, pictures, faces, smells.

      Benefits and Military Significance Understanding the relationship between exposure to repetitive, sub-concussive impacts to behavioural symptomatology, vestibular ocular dysfunction, brain electrophysiology, and cognition to aid in early detection/prevention, treatment and prognostication of SOF members. Moreover, this study will lay the foundation for future research for years to come.

ELIGIBILITY:
Inclusion Criteria:

* ● Male or female between 18 and 65

  * Normal or corrected to normal vision and hearing (Note: If the patient has hearing aids or wears glasses, they are still able to complete the assessment. They will need to remove hearing aids for the Attention & Concentration and Information Processing test)
  * Sit still for 10-15 minutes
  * Understand basic instructions of cognitive tests

Exclusion Criteria:

* ● Metal plates under their scalp that cross the midline

  * Taking epilepsy medications
  * History of neurologic or neuropsychiatric disorder prior to concussion in controls
  * Taking psychotropic medications
  * History of complete deafness
  * Supplements or performance enhancing drugs that can affect brain function

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — man, woman and other
Study Population: A sample will be recruited from a group of 20 CAF SOF personnel ages 18-65 will be assessed twice: pre and post-special forces military training. All members enrolled in this training will be invited to participate in the study. Testing periods will be about 4 weeks apart, with post training testing within 1 week of conclusion of the exercise. Patients will be recruited from within the Canadian Special Operation Forces community
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Event Related Potential Changes | baseline and within 1 week of completion of 4 week training course
  changes on selected event related potentials (ie N100, P200, N200, P300, N400) when testing attention, concentration, continuous visual memory, executive function and comprehension

SECONDARY OUTCOMES:
Impact Cognitive testing | baseline and within 1 week of completion of 4 week training course
  FDA cleared online tool for baseline and post-injury testing. It measures patient reported symptoms, visual and verbal memory, reaction time, and processing speed to help determine if a patient can safely return to activity.
VOMS | baseline and within 1 week of completion of 4 week training course
  Vestibular Ocular Motor Screening (VOMS) consists of symptom reporting (eg headache, dizziness, nausea, and fogginess) ranging from 0 (none) to 10 (severe) after testing smooth pursuits, saccades (horizontal and vertical), convergence, Neer Point of Convergence (NPC) distance, horizontal VOR, vertical VOR, and visual motor sensitivity (VMS). For the purpose of this study, we will use the VOMS cutoff scores of ≥2 total symptom score on any VOMS subscale and/or ≥5 cm on NPC average distance

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, Principal Investigator — Gaurav Gupta MPC
Locations (1):
- Canadian Forces Health Services, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No